CLINICAL TRIAL: NCT03269526
Title: Phase Ib/II Treatment of Advanced Pancreatic Cancer With Anti-CD3 x Anti-EGFR-Bispecific Antibody Armed Activated T-Cells (BATs)
Brief Title: BATs Treatment for Pancreatic Cancer, Phase Ib/II
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Tri Minh Le, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19236
Record Dates: First submitted 2017-08-11; First posted 2017-08-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; Pancreatic Adenocarcinoma; Adoptive cell therapy; Armed activated T-cells; Bispecific antibody; Immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Standard of care chemotherapy followed by Anti-CD3 x anti-EGFR-Bispecific Antibody Armed Activated T-cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGFR BATs after standard of care chemo (Experimental): Subjects will undergo apheresis to collect peripheral blood mononuclear cells. Cells will be cultured for up to 2 weeks before activated T-cells will be harvested, armed with EGFR Biarmed activated T-cells, washed to remove unbound EGFRBi, and cryopreserved. Subjects will then receive one dose of standard of care chemotherapy prior to receiving EGFR BATs.
  Interventions: Drug: EGFR BATs after standard of care chemo

INTERVENTIONS:
Drug: EGFR BATs after standard of care chemo — Subjects will receive one dose of standard of care chemotherapy prior to twice weekly or weekly infusions of EGFR BATs for 4 weeks.

SUMMARY:
This protocol will confirm toxicities and estimate the clinical efficacy of combining anti-CD3 x anti-EGFR bispecific antibody (EGFRBi) armed activated T cells (EGFR BATs) given to patients with locally advanced or metastatic pancreatic cancer who have received at least one dose of first line chemotherapy and may have responding, stable or progressive disease. Phase Ib will confirm a safe dose of 8 infusions, given twice weekly, of EGFR-BATs in 3 to 6 subjects. The phase II portion of the trial will test the clinical efficacy of this dose in 22 patients (including those in Phase Ib).

DETAILED DESCRIPTION:
Once subjects are determined eligible, white blood cells (lymphocytes) are collected via leukapheresis procedure at approximately 3 to 4 weeks prior to first EGFR-BATs infusion. The white blood cells, specifically T cells, are then mixed with two proteins - OKT3 and IL-2 which activates the cells to multiply. After approximately 14 days in culture, the activated T cells are coated with the OKT3 and cetuximab to produce bispecific antibody armed T cells (BATs). Cells are then frozen and stored until scheduled to be infused.

Within one to two weeks prior to infusion of the study treatment, subjects will receive one dose of chemotherapy. The choice of chemotherapy agent(s) is at the discretion of the treating physician.

At approximately 4 weeks following leukapheresis procedure, twice weekly or weekly infusions of the BATs cells will take place (twice weekly for participants enrolled before DATE and weekly for participants enrolled after DATE). A total of eight twice weekly infusions or four weekly infusions will be given over a four week period. Please note that the weekly dose for both groups of participants is the same; participants that received twice weekly dosing received half of the weekly dose at each infusion.

Follow-up appointment schedule will include clinic visits at 1 to 2 weeks, 4 to 5 weeks, 2 months, 4 months and 6 months following the last infusion of BATs cells.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of pancreatic adenocarcinoma. Must have locally advanced or metastatic pancreatic cancer and received at least one dose of chemotherapy (any treatment line) and may have responding, stable or progressive disease
2. Expected survival ≥ 3 months
3. ECOG Performance Status 0 or 1
4. Left Ventricular Ejection Fraction (LVEF) ≥ 45% at rest (MUGA or Echo)
5. Age ≥ 18 years at the time of consent (Written informed consent and HIPAA authorization for release of personal health information)
6. Females of childbearing potential, and males, must be willing to use an effective method of contraception
7. Females of childbearing potential must have a negative pregnancy test within 10 days prior to "on study" status. If a urine or serum test is positive or cannot be confirmed as negative, the other (urine or serum pregnancy test, whichever was not performed first) will be required.
8. Demonstrate adequate hepatic, renal, and bone marrow function as defined below; all hematological, renal, and hepatic screening labs should be performed within 10 days prior to "on study" status (alpha gal testing must be within the regular screening period).

   * Absolute lymphocyte count ≥ 400/mm3
   * Absolute neutrophil count (ANC) ≥ 1,000/mm3
   * Platelets ≥ 75,000/mm3
   * Hemoglobin ≥ 8 g/dL
   * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) < 2.0 mg/dl OR ≥50 ml/mm
   * Serum total bilirubin ≤ 2 mg/dl (biliary stent is allowed)
   * AST (SGOT) and ALT (SGPT) < 5.0 times normal
   * Alpha 1,3 Galactose IgE ("alpha gal") < 0.35 IU/ml or "negative"

Exclusion Criteria:

1. Known hypersensitivity to cetuximab or other EGFR antibody
2. Treatment with any investigational agent within 14 days prior to first study intervention (apheresis) for protocol therapy
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to first study intervention (apheresis). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
4. Serious non-healing wound, ulcer, bone fracture, major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to "on-study" status
5. Active liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
6. Is HIV positive or has evidence of active Hepatitis C virus or active Hepatitis B virus. If initial Hepatitis C test shows a positive result, the patient should have a Hepatitis viral load test to confirm. If initial HIV or Hepatitis B virus testing shows a positive result, no further testing will be done.
7. Active bleeding or a pathological condition that is associated with a high risk of bleeding (therapeutic anticoagulation is allowed)
8. Has an active infection requiring systemic therapy
9. A serious uncontrolled medical disorder that in the opinion of the Investigator may be jeopardized by the treatment with protocol therapy
10. Has a known history of active TB (Bacillus Tuberculosis)
11. Has had prior chemotherapy, radiation, hormonal, monoclonal antibody (mAb) or targeted small molecule therapy, within 2 weeks prior to the first study procedure (apheresis). Subjects who have not recovered to <Grade 3 from an adverse event due to a previously administered agent are not eligible.
12. Has received a live vaccine within 30 days of first study procedure (apheresis).
13. History of a recent myocardial infarction (within one year), a past myocardial infarction (more than one year ago) along with current coronary symptoms requiring medications.
14. Has history of another malignancy within the past 5 years. Exceptions include

    * basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy
    * in situ cervical cancer.
15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Females must not be breastfeeding
18. Pt may be excluded if, in the opinion of the PI and investigator team, the pt is not capable of being compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From the beginning of treatment (bridging chemotherapy) until no sooner than 30 days following the last study treatment
  Safety will be assessed by incidence and severity of adverse events, changes in laboratory findings, physical examinations, vital signs, and the number of dose limiting toxicities and other discontinuations due to adverse events.
Overall survival | Until subject's death or study closure (whichever occurs first) for an average of 36 months from study treatment completion
  An improvement in median overall survival (OS), defined as an increase from historical data of 8.7 months to 18.0 months.

SECONDARY OUTCOMES:
Cellular or humoral anti-pancreatic cancer responses | Every 2-6 months after the last EGFR BATs infusion for as long as the response lasts -- an average of 4 months
  These will be measured in peripheral blood mononuclear cells
Clinical Efficacy | Imaging will be performed prior to treatment, 2 months after the last BATs infusion, then according to standard of care for an average of 12 months
  Progression-free survival, measured by immune-related response criteria (irRC)
Examine tumor tissue for immune system cells, cytokines and proteins to estimate whether the type and number of immune cells correlates with clinical responses | Tumor paraffin blocks from tissue collected prior to treatment will be batched and analyzed within 1 year of completion of study accrual
  These immune system cells, cytokines and proteins include CD3, CD4, CD8, PD1/PDL1, monocytes subpopulations, MDSCs, and cytoplasmic IFN-y, tumor infiltrating lymphocytes, and IL-10. This will be measured using immunohistochemical staining to quantitate type and number of immune system cells, cytokines, and proteins to estimate whether the type and number correlate with clinical responses.

CONTACTS AND LOCATIONS:
Overall Officials: Tri Le, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum LG, Thakur A, Al-Kadhimi Z, Colvin GA, Cummings FJ, Legare RD, Dizon DS, Kouttab N, Maizel A, Colaiace W, Liu Q, Rathore R. Targeted T-cell Therapy in Stage IV Breast Cancer: A Phase I Clinical Trial. Clin Cancer Res. 2015 May 15;21(10):2305-14. doi: 10.1158/1078-0432.CCR-14-2280. Epub 2015 Feb 16. PMID 25688159
- [Background] Vaishampayan U, Thakur A, Rathore R, Kouttab N, Lum LG. Phase I Study of Anti-CD3 x Anti-Her2 Bispecific Antibody in Metastatic Castrate Resistant Prostate Cancer Patients. Prostate Cancer. 2015;2015:285193. doi: 10.1155/2015/285193. Epub 2015 Feb 23. PMID 25802762